CLINICAL TRIAL: NCT03145896
Title: The Correlation Between Anemia of Chronic Diseases, Hepcidin and Vitamin D in IBD Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, michal roll, Phd, Tel-Aviv Sourasky Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TASMC-15-SC-0778-CTIL
Record Dates: First submitted 2017-04-05; First posted 2017-05-09 (Actual); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: IBD
Keywords: vitamin D; Anemia; IBD
MeSH Terms: conditions — Anemia | interventions — Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IBD patients with Vitamin D treatment (Active Comparator)
  Interventions: Dietary Supplement: vitamin D
- IBD patients with no Vitamin D treatment (No Intervention)

INTERVENTIONS:
Dietary Supplement: vitamin D — After the gastroscopy all patients will be taught to take 4000 unit of vitamin D (25(OH)D) daily (not a specific brand) , for the next 2 week. All patients will be invited for follow-up in 2 weeks to get the histopathology result. In this encounter we will take again blood sample for 25(OH)D, calcium, phosphate, CRP and complete blood count including hemoglobin. a control group will not take the Vitamin D supplements.
  Arms: IBD patients with Vitamin D treatment

SUMMARY:
Crohn's disease (CD) and ulcerative colitis (UC) are chronic gastrointestinal diseases characterized by relapsing and remitting inflammation of the intestines Anemia may often complicate the course of inflammatory bowel disease (IBD). The cause of anemia in IBD is multifactorial In the chronically ill patients, it has been described that the mechanism underlying anemia involves hepcidin.A potential mechanism underlying anemia during an chronic disease is suggested by recent data demonstrating a hepcidin lowering effect of vitamin D

DETAILED DESCRIPTION:
Crohn's disease (CD) and ulcerative colitis (UC) are chronic gastrointestinal diseases characterized by relapsing and remitting inflammation of the intestines . Anemia may often complicate the course of inflammatory bowel disease (IBD) . A recent systematic review showed that anemia is common and may affect roughly 17% of patients with IBD .

The cause of anemia in IBD is multifactorial. The most common cause for anemia in IBD patients is iron deficiency anemia (IDA) secondary to increased blood loss from inflamed gastrointestinal mucosa and impaired absorption of iron. The anemia can be macrocytic due to impaired absorption of other nutrients including folate and cobalamin. Other causes are anemia due to medication (such as sulfasalazine) and anemia of chronic disease (ACD) .

ACD is characterized by normochromic, normocytic or mildly microcytic erythrocytes, low or normal serum iron and total iron-binding capacity, normal or increased iron stores reflected by elevated ferritin levels, low transferrin levels, and an inappropriately low reticulocyte response relative to the degree of anemia. ACD is unresponsive to treatment with iron, vitamin B12 or folic acid.

In the chronically ill patients, it has been described that the mechanism underlying anemia involves hepcidin.

Hepcidin, a β-defensin-like antimicrobial peptide, is part of the innate immune system and thus constitutes the first-line defense against infections. In vivo and in vitro studies have demonstrated that hepcidin is active against Gram-positive and Gram-negative bacteria as well as yeasts . In addition to its antimicrobial activity, it acts as an iron regulatory hormone. Increased hepcidin synthesis inhibits iron flow into plasma from macrophages that have taken up and degraded senescent erythrocytes as well as their hemoglobin, and also from small intestinal epithelial cells involved in the absorption of dietary iron . This iron release from cytoplasmic stores is prevented by binding of hepcidin to the iron exporter protein ferroportin. Ferroportin is internalized and degraded upon hepcidin activity.

Hepcidin is produced and secreted mainly by hepatocytes, and to a lesser extent by macrophages and adipocytes . Its synthesis is regulated by iron, erythropoietic activity and inflammation . Hepcidin expression is down-regulated in anemia with concomitant iron deficiency. Thus, ferroportin is not internalized from the cell membrane and iron can be transported from stores to the plasma to provide heme synthesis and erythropoiesis with more iron. On the other hand during anemia of chronic diseases (without significant iron deficiency), hepcidin expression is even increased, which may explain why iron is "trapped" intracellularly under these conditions.

In IBD (similar to other chronic inflammatory disease or infections), it can be assumed that inflammation increases hepcidin expression and synthesis as hepcidin also is an "acute phase protein" . This induction of hepcidin protein synthesis is at least partially mediated by interleukin-6 via its receptor and subsequent intracellular signal transduction via signal transducer and activator of transcription-3 (STAT3).

In the study of Pantelis et el it was found that the median hepcidin level were significantly higher in patients with IBD compared with healthy controls In a recent study by Basseri and coworkers, a positive correlation between serum hepcidin and IL-6 levels in IBD patients was confirmed. The authors further detected a negative correlation between serum hepcidin concentration and Hgb levels.

A potential mechanism underlying anemia during an chronic disease is suggested by recent data demonstrating a hepcidin lowering effect of vitamin D.

In the setting of chronic kidney disease patients, it was shown that vitamin D is inversely associated with hepcidin concentrations, and positively associated with hemoglobin and iron concentrations. Importantly, vitamin D has been reported to decrease inflammatory cytokines implicated in the pathophysiology of anemia during inflammation, and suppress expression of hepcidin mRNA. Additionally, oral administration of vitamin D in healthy adult volunteers lowered serum levels of hepcidin by 50% compared to baseline levels within 24 hours and persisted for 72 hours.

These initial results seem promising; but thus far the association between IBD, vitamin D status and anemia has never been established in the pediatric population, nor has the connection between these hormones and the efficacy of iron supplementation therapy. Controlled studies are warranted to determine this link and, thereafter, investigate the possible therapeutic potential of vitamin D supplementation

Aim:

To examine the association between hepcidin, IL6, vitamin D and anemia in children and adolescence with IBD and to study the possible effect of vitamin D supplementation on hepcidin level in IBD patients.

Hypothesis:

We hypothesize that in patients with parameters of anemia of chronic disease hepcidine level will be high and vitamin D level will be low. Supplementation of vitamin D will lower hepcidin levels and improve the anemia.

Study population and study design:

This is a prospective study. It will take place in the Pediatric Gastroenterology Unit at Dana- Dwek Children's hospital.

The study population will consists of 40 newly diagnosed IBD Patients, male and female, age 6-18. We will recruit all patients that are suspicious to have IBD based on their clinical and laboratory evaluation in their first diagnostic colonoscopy.

Each participant in the study will provide written informed consent at the beginning of the study.

We will document the participant's age, sex, anthropometric measurements (weight, height).

Each participant will complete a questionnaire that records personal lifestyle and demographic information, physical activity and sun exposure. Medical data (medical background, medication, sign and symptoms, severity of disease) will be collected from the patient's medical file.

We will take from each participant blood sample (approximately 10cc), to test levels of 25(OH)D, calcium, phosphate, CRP and complete blood count including hemoglobin, hematocrit (Hct), RBC, MCV, RDW, serum iron, total-iron-binding capacity, hepcidin, transferrin, soulable transferrin receptor, ferritin and IL6. We will document calprotectin level if available.

Before discharge home all patients will be taught to take 5000 unit of vitamin D (25(OH)D) daily, for the next 2 week . All patients will be invited for follow-up in 2 weeks to get the histopathology result. In this encounter we will take again blood sample for 25(OH)D, calcium, phosphate, CRP and complete blood count including hemoglobin, hematocrit (Hct), RBC, MCV, RDW, serum iron, total-iron-binding capacity, hepcidin, transferrin, ferritin soulable transferrin receptor and IL6.

All the data will be coded and the questionnaires will be kept in a locked place.

The concentration of 25(OH)D will be measured by radioimmunoassay. Levels of Hepcidin will be measured by a commercial kit.

Blood sample collection and questionnaire completion will be done in 2 days. (Visits will be appointed as the usual appointments after endoscopy in our clinic).

Study data analysis will be completed within a year.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed IBD based on histopathology.

Exclusion Criteria:

* Patients that their histopathology will confirm eventually different diagnosis.
* Participants that are receiving medications known to alter vitamin D metabolism or have hepatic or renal disease
* Participants that suffer from hemoglobinopaties, bone marrow failure, or receive bone marrow suppressing agents
* Participants that went through a recent surgical procedure, or needed blood transfusion for any reason

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-06-01 (Estimated); Primary Completion 2018-06-01 (Estimated); Study Completion 2018-09-01 (Estimated)

PRIMARY OUTCOMES:
influence of vitamin D on anemia of inflammation | 2 weeks
  levels of hepcidin, IL6, vitamin D and anemia in children and adolescence with newly diagnosed IBD before and after vitamin D supplemntation.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Podolsky DK. Inflammatory bowel disease. N Engl J Med. 2002 Aug 8;347(6):417-29. doi: 10.1056/NEJMra020831. No abstract available. PMID 12167685
- [Background] Gasche C. Anemia in IBD: the overlooked villain. Inflamm Bowel Dis. 2000 May;6(2):142-150; discussion 151. doi: 10.1097/00054725-200005000-00013. PMID 10833075
- [Background] de la Morena F, Gisbert JP. [Anemia and inflammatory bowel disease]. Rev Esp Enferm Dig. 2008 May;100(5):285-93. Spanish. PMID 18662081
- [Background] de Silva AD, Mylonaki M, Rampton DS. Oral iron therapy in inflammatory bowel disease: usage, tolerance, and efficacy. Inflamm Bowel Dis. 2003 Sep;9(5):316-20. doi: 10.1097/00054725-200309000-00005. PMID 14555915
- [Background] Gisbert JP, Gomollon F. Common misconceptions in the diagnosis and management of anemia in inflammatory bowel disease. Am J Gastroenterol. 2008 May;103(5):1299-307. doi: 10.1111/j.1572-0241.2008.01846.x. PMID 18477354
- [Background] Basseri RJ, Nemeth E, Vassilaki ME, Basseri B, Enayati P, Shaye O, Bourikas LA, Ganz T, Papadakis KA. Hepcidin is a key mediator of anemia of inflammation in Crohn's disease. J Crohns Colitis. 2013 Sep;7(8):e286-91. doi: 10.1016/j.crohns.2012.10.013. Epub 2012 Dec 6. PMID 23219355
- [Background] Yapakci E, Tarcan A, Celik B, Ozbek N, Gurakan B. Serum pro-hepcidin levels in term and preterm newborns with sepsis. Pediatr Int. 2009 Apr;51(2):289-92. doi: 10.1111/j.1442-200X.2008.02688.x. PMID 19405934
- [Background] Nemeth E, Ganz T. The role of hepcidin in iron metabolism. Acta Haematol. 2009;122(2-3):78-86. doi: 10.1159/000243791. Epub 2009 Nov 10. PMID 19907144
- [Background] Ruchala P, Nemeth E. The pathophysiology and pharmacology of hepcidin. Trends Pharmacol Sci. 2014 Mar;35(3):155-61. doi: 10.1016/j.tips.2014.01.004. Epub 2014 Feb 17. PMID 24552640
- [Background] Ross SL, Tran L, Winters A, Lee KJ, Plewa C, Foltz I, King C, Miranda LP, Allen J, Beckman H, Cooke KS, Moody G, Sasu BJ, Nemeth E, Ganz T, Molineux G, Arvedson TL. Molecular mechanism of hepcidin-mediated ferroportin internalization requires ferroportin lysines, not tyrosines or JAK-STAT. Cell Metab. 2012 Jun 6;15(6):905-17. doi: 10.1016/j.cmet.2012.03.017. PMID 22682226
- [Background] Dudkowiak R, Neubauer K, Poniewierka E. Hepcidin and its role in inflammatory bowel disease. Adv Clin Exp Med. 2013 Jul-Aug;22(4):585-91. PMID 23986220
- [Background] Nemeth E, Valore EV, Territo M, Schiller G, Lichtenstein A, Ganz T. Hepcidin, a putative mediator of anemia of inflammation, is a type II acute-phase protein. Blood. 2003 Apr 1;101(7):2461-3. doi: 10.1182/blood-2002-10-3235. Epub 2002 Nov 14. PMID 12433676
- [Background] Theurl I, Schroll A, Nairz M, Seifert M, Theurl M, Sonnweber T, Kulaksiz H, Weiss G. Pathways for the regulation of hepcidin expression in anemia of chronic disease and iron deficiency anemia in vivo. Haematologica. 2011 Dec;96(12):1761-9. doi: 10.3324/haematol.2011.048926. Epub 2011 Aug 22. PMID 21859731
- [Background] Ferrucci L, Semba RD, Guralnik JM, Ershler WB, Bandinelli S, Patel KV, Sun K, Woodman RC, Andrews NC, Cotter RJ, Ganz T, Nemeth E, Longo DL. Proinflammatory state, hepcidin, and anemia in older persons. Blood. 2010 May 6;115(18):3810-6. doi: 10.1182/blood-2009-02-201087. Epub 2010 Jan 15. PMID 20081092
- [Background] Nemeth E, Rivera S, Gabayan V, Keller C, Taudorf S, Pedersen BK, Ganz T. IL-6 mediates hypoferremia of inflammation by inducing the synthesis of the iron regulatory hormone hepcidin. J Clin Invest. 2004 May;113(9):1271-6. doi: 10.1172/JCI20945. PMID 15124018
- [Background] Oustamanolakis P, Koutroubakis IE, Messaritakis I, Malliaraki N, Sfiridaki A, Kouroumalis EA. Serum hepcidin and prohepcidin concentrations in inflammatory bowel disease. Eur J Gastroenterol Hepatol. 2011 Mar;23(3):262-8. doi: 10.1097/MEG.0b013e328343b885. PMID 21285884
- [Background] Smith EM, Alvarez JA, Martin GS, Zughaier SM, Ziegler TR, Tangpricha V. Vitamin D deficiency is associated with anaemia among African Americans in a US cohort. Br J Nutr. 2015 Jun 14;113(11):1732-40. doi: 10.1017/S0007114515000999. Epub 2015 Apr 16. PMID 25876674
- [Background] Bacchetta J, Zaritsky JJ, Sea JL, Chun RF, Lisse TS, Zavala K, Nayak A, Wesseling-Perry K, Westerman M, Hollis BW, Salusky IB, Hewison M. Suppression of iron-regulatory hepcidin by vitamin D. J Am Soc Nephrol. 2014 Mar;25(3):564-72. doi: 10.1681/ASN.2013040355. Epub 2013 Nov 7. PMID 24204002
- [Derived] Moran-Lev H, Galai T, Yerushalmy-Feler A, Weisman Y, Anafy A, Deutsch V, Cipok M, Lubetzky R, Cohen S. Vitamin D Decreases Hepcidin and Inflammatory Markers in Newly Diagnosed Inflammatory Bowel Disease Paediatric Patients: A Prospective Study. J Crohns Colitis. 2019 Sep 27;13(10):1287-1291. doi: 10.1093/ecco-jcc/jjz056. PMID 30840757